CLINICAL TRIAL: NCT04518891
Title: Efficacy of the Cognitive Functional Therapy (CFT) in Patients With Chronic Nonspecific Low Back Pain: a Study Protocol for a Randomized Sham-controlled Trial
Brief Title: Cognitive Functional Therapy Compared With Sham-treatment for Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Thais Cristina Chaves, Director, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2604/2020
Record Dates: First submitted 2020-08-15; First posted 2020-08-19 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Chronic Low-back Pain
Keywords: Cognitive Functional Therapy; Low Back Pain; Pain Management; Placebo Effect; Self-efficacy
MeSH Terms: conditions — Low Back Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Functional Therapy (CFT) Group (Experimental): There will be 3 main components in the intervention:
  1. Making sense of pain: the cognitive component will focus on identifying the factors that contribute to pain during examination. This will include discussion on the multidimensional nature of persistent pain, individual beliefs, and how emotions and behaviours regarding movement and lifestyle can reinforce a vicious cycle of pain and disability.
  2. Controlled exposure: specific functional training is designed to normalise maladaptive or provocative movement and posture. functional integration is directed at activities of daily life that are avoided by the patient. This will vary among individuals but should include basic activities such as rolling in bed, sitting, sitting to standing, walking, bending and lifting.
  3. Lifestyle change: Physical activity and lifestyle. Patients will be advised to gradually increase physical activity based on their preference, while also focusing on sleep hygiene, stress and management strategies.
  Interventions: Behavioral: Cognitive Functional Therapy (CFT)
- Sham intervention (Sham Comparator): Placebo group will be treated with detuned photobiomodulation device (904Nm Ibramed Infrared - no-visible beam), without any emission of therapeutic dose. Nine sites will be applicate on the patient's lumbar region: three central sites on top of the spinous processes (between T11 and T12, L2 and L3, L5 and S1); in the same direction, but laterally, three sites on the left and three on the right. Three minutes of fake stimulation will be administered, summing up 27 minutes. In addition, a neutral talking control therapy of at least 15 minutes will be provided to patients in each session. Maladaptive beliefs will not be challenged; however, the therapists will be trained to show interest and warmth, empathy and encouraging participants to discuss neutral topics such as hobbies, sports, and current affairs. No advice or problem solving will be given, and any attempt to talk about emotional issues will be kindly discouraged and the talking will be redirect to neutral tropics.
  Interventions: Device: Sham intervention

INTERVENTIONS:
Behavioral: Cognitive Functional Therapy (CFT) — Cognitive functional therapy (CFT) is an intervention that deals with potentially modifiable multidimensional aspects of pain (e.g. provocative cognitive, movement and lifestyle behaviours). Treatment with CFT will be individualised, the physiotherapist will listen to the complete patient pain history and the intervention will be focused on individual needs. A detailed examination will be crucial in identifying the modifiable multidimensional mediators of pain and disability (provocative cognitive, pain, movement and lifestyle behaviors) of each participant.
  Arms: Cognitive Functional Therapy (CFT) Group
Device: Sham intervention — Due to the impossibility of applying placebo exercise, the control intervention in this study will be based on successful reports of placebo intervention in patients with chronic low back pain in the literature (Placebo photobiomodulation + neutral talking control)
  Other Names: Placebo photobiomodulation + neutral listening
  Arms: Sham intervention

SUMMARY:
Chronic low back pain is a public health problem, and there is strong evidence that it is associated with a complex interaction of biopsychosocial factors. Cognitive functional therapy (CFT) is a promising new intervention that deals with potentially modifiable multidimensional aspects of pain (eg, provocative cognitive, movement and lifestyle behaviors). In order to better understand the contextual effects, the aim of the current study is to investigate the efficacy of CFT compared with a sham-intervention for pain intensity and disability post-intervention in patients with non-specific chronic low back pain (CLBP).

This study is a randomized clinical trial (RCT) in which 152 (18 - 60 years old) patients with CLBP will be enrolled. The patients will be randomly allocated to receive: (1) CFT intervention or (2) sham-intervention. The experimental group will receive individualized CFT in a pragmatic manner (5 to 7 sessions) based on the clinical progression of participants. The sham group will attend six sessions: consisted of 30 minutes of photobiomodulation using a detuned device and more 15 minutes of talking about neutral topics. Participants will be assessed pre and post-intervention, three months and six months after randomization. Patients from both groups also will receive an educational booklet. The primary outcomes will be pain intensity and disability post-intervention. The secondary outcomes will be: pain intensity and disability at 3- and 6-month follow-up, as well as self-efficacy, global perceived effect of improvement and functioning post-intervention, 3- and 6-month follow-up. The patients and the assessor will be blinded to treatment administered (active vs. sham).

The between-group differences (effects of treatment) and their respective 95% confidence intervals will be calculated by constructing linear mixed models. Treatment effect for the primary and secondary outcomes will be estimated using mixed linear models.

To the best of our knowledge, the current study will be the first to compare CFT vs. sham intervention. Sham-controlled RCTs may help to understand the influence of non-specific factors on treatment outcomes. Considering complex interventions as CFT, it is imperative to understand the impact of contextual factors on outcomes.

DETAILED DESCRIPTION:
The aim of the current study is to investigate the efficacy of Cognitive Functional Therapy (CFT) compared with a sham-intervention (sham photobiomodulation + neutral talking), for pain intensity and disability post-intervention in patients with non-specific chronic low back pain (CLBP). The secondary aims will be to investigate the effect of CFT for pain intensity and disability at 3- and 6-month follow-up, as well as the effect of the active treatment on self-efficacy, global perceived effect of improvement and functioning post-intervention, 3- and 6-month follow-up.

The study was submitted to and approved by the ethics committee for research involving human subjects of the Ribeirão Preto Medical School (Ethics Committee Board from Centro Saúde Escola Cuaibá) of the University of São Paulo (HCFMRP CAE number: 26780619.0.0000.5414). Written informed consent will be obtained from all participants included in the study. No significant adverse reactions are anticipated in the study, but these will be monitored.

This study will be a sham-controlled RCT and will follow the recommendations described on Consolidated Standards of Reporting Trials (CONSORT) statement. The sample will be comprised of 152 participants (both genders) with non-specific CLBP who will be referred to the physiotherapy outpatient clinic from Ribeirão Preto Medical School - University of São Paulo (Brazil).

Patients will be informed that this study will involve a sham intervention arm (fake intervention in which an inert treatment will be provided but it still can result in positive outcomes due to its psychological effects) vs. an active treatment arm, but the nature of the sham will not be elucidated (equipment detuned).

After this initial assessment, participants will be randomly assigned using block randomization by simple computerized procedures to one of the two treatment groups through the use of cards previously placed in opaque sealed envelopes: i) CFT group or ii) Sham group.

As a strategy to control for the treatment fidelity on both arms of the study, we will adopt the framework developed by the NIH Behaviour Change Consortium (BCC). To control for the "Intervention Delivery", the time of therapist-patient interaction, number of sessions and the different components of the intervention administered (e.g.: in the sham-group, the time administering the sham photobiomodulation and the time spent with neutral talking), as well as video recordings along the trial will be registered. Also, regular meetings to discuss the clinical cases will be performed. Furthermore, the "Intervention receipt" will be assessed in two different manners: i) on the completion of the study, each participant will be submitted to a manipulation check and they will be asked about the group they think they were at and ii) patients in both groups will be invited to summarize at the beginning of each session how the treatment impact their lives.

Despite it is a sham-controlled RCT, considering the differences in the interventions administered in both study arms, it will not be possible to blind the therapists, however, patients will be blinded to randomized interventions. The assessor and the participants will not have access to what type of treatment the participant will be given.

To the best of our knowledge, the current study will be the first to compare CFT vs. sham intervention. Sham-controlled RCTs may help to understand the influence of non-specific factors on treatment outcomes. Considering complex interventions as CFT, it is imperative to understand the impact of contextual factors on outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 60 years;
* Current episode of CLBP lasting more than 3 months (including cases with pain in the lower limbs);
* Seeking primary clinical care for at least 6 weeks ago for this episode of low back pain;
* Primary pain located between T12 and the gluteal folds;
* Pain intensity equal to or greater than 4 on the 0-10 numerical pain scale;
* Pain caused by certain postures, activities and movements;
* Score greater than 14% on the Oswestry Disability Index;
* And be able to speak and understand Portuguese well to complete the questionnaires.

Exclusion Criteria:

* Classification in red flags (neoplastic diseases or tumors in the spine, inflammatory diseases, infections and fractures);
* Leg pain as a primary problem (eg nerve root compression or disc prolapse with active radiculopathy, or lumbar stenosis);
* Previous physiotherapy treatments (less than six months before the evaluation period);
* History of spine surgery;
* Pregnancy;
* Rheumatological / inflammatory disease;
* Progressive neurological disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 152 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity: Numeric pain rating scale (NPRS) | Post-intervention
  The NPRS used in this trial will consist of numbers from 0 to 10, in which 0 represents "no pain" and 10 represents "worst pain imaginable". High scores mean worse pain intensity.
Low Back Pain Related Disability: Oswestry Disability Index (ODI) | Post-intervention
  The ODI consists of 10 items, each of which has six response options. The total score will be calculated by summing up all the points, ranging from 10 to 50. This sum will be transformed into a percentage (0 to 100). High scores mean worse disability.

SECONDARY OUTCOMES:
Pain intensity: Numeric pain rating scale (NPRS) | 3 and 6 months after randomization
  The NPRS used in this trial will consist of numbers from 0 to 10, in which 0 represents "no pain" and 10 represents "worst pain imaginable". High scores mean worse pain intensity.
Low Back Pain Related Disability: Oswestry Disability Index (ODI) | 3 and 6 months after randomization
  The ODI consists of 10 items, each of which has six response options. The total score will be calculated by summing up all the points, ranging from 10 to 50. This sum will be transformed into a percentage (0 to 100). High scores mean worse disability.
Pain Self-Efficacy: Pain Self-Efficacy Questionnaire (PSEQ) | Post-intervention, 3 and 6 months after randomization
  The PSEQ has 10 items related individual's confidence to perform a certain task which are rated on a 7-point ordinal scale (ranging from 0: "not at all confident" to 6: "completely confident"). The score ranges from 0 to 60, higher score means better self-efficacy.
Global perceived effect: Global Perceived Effect Scale (GPES) | Post-intervention, 3 and 6 months after randomization
  GPES is an 11-point scale ranging from -5 ("vastly worse") through 0 (no change) to +5 (completely recovered).Higher score means better perception of improvement.
Function: Patient Specific Functional Scale (PSFS) | Post-intervention, 3 and 6 months after randomization
  In the PSFS patients are asked to identify up to three important activities that they are having difficulties with or are unable to perform due to their condition. In addition, the patients are asked to rate, on an 11-point scale (ranging from 0 to 10) their current level of ability associated with each activity. Score ranges from 0 (unable to perform) to 10 (able to perform at preinjury level). Higher score means better function.

OTHER OUTCOMES:
Expactation: Standford ExpectationTreatment Scale (SETS) | Baseline
  The SETS is a scale with six items, three covering positive treatment related expectations and three regarding negative treatment related expectations. The SETS is comprised of a seven-point Likert-type response scale was chosen, varying from (1) 'strongly disagree' to (7) 'strongly agree'. An average of items 1, 3, and 5 yields the positive expectancy score (higher score means strong positive expectation), while an average of 2, 4, and 6 yields the negative expectancy score (higher score means strong negative expectation).
Depression: Patient Health Questionnaire 9-item (PHQ-9) | Baseline
  The PHQ-9 is a nine-item questionnaire designed to screen for depression in primary care and other medical settings. They incorporate DSM-IV depression criteria with other leading major depressive symptoms into a brief self-report instrument. Score ranges from 0 to 21. The standard cut-off score for screening to identify possible major depression is 10 or above.
Anxiety: Generalized Anxiety Disorder 7-item scale (GAD7) | Baseline
  The GAD-7 is a 7-item self-report measure of generalized anxiety symptoms grouped into one factor of generalized anxiety. Respondents score each item in a 4-point scale based on how often they have been bothered by the described symptoms over the last two weeks (not at all = 0; several days = 1; more than half the days = 2; nearly every day = 3). Total scores range from 0 to 21, with higher scores reflecting higher severity levels of anxiety.
Kinesiophobia: Tampa Scale for Kinesiophobia (TSK) | Baseline
  This scale was used to assess fear and avoidance beliefs about movement and reinjury. The 17 statements were scored on 4-point scales from ''strongly disagree'' to ''strongly agree,'' yielding a total range from 17 to 68. Higher scores indicate more severe fear-avoidance beliefs.
Catastrophizing: Pain Catastrophizing Scale (PCS) | Baseline
  The scale is composed of 13 items, the total score is the sum of the items divided by the number of items answered, with the minimum score being 0 and the maximum being 5 for each item. Higher scores indicated a greater presence of catastrophic thoughts.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana R Lira, Master, Principal Investigator; Ney A Meziat, PhD, Study Director — Augusto Motta University Center (UNISUAM); Thais C Chaves, PhD, Study Director — University of Sao Paulo
Locations (1):
- University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Lira MR, Meziat-Filho N, Zuelli Martins Silva G, Castro J, Fernandez J, Guirro RRJ, Berg R, Chaves TC. Efficacy of cognitive functional therapy for pain intensity and disability in patients with non-specific chronic low back pain: a randomised sham-controlled trial. Br J Sports Med. 2025 Jun 18;59(13):912-920. doi: 10.1136/bjsports-2024-109012. PMID 40049758
- [Derived] de Lira MR, de Mello Meziat-Filho NA, Silva GZM, Chaves TC. Efficacy of the cognitive functional therapy (CFT) in patients with chronic nonspecific low back pain: a study protocol for a randomized sham-controlled trial. Trials. 2022 Jul 4;23(1):544. doi: 10.1186/s13063-022-06466-8. PMID 35788240